CLINICAL TRIAL: NCT07232251
Title: Evaluation of the Effects of Different Intraoperative Warming Techniques on Core Body Temperature and Hematologic Inflammatory Indices (SII, NLR, PLR, LMR) in Patients Undergoing Laparoscopic Cholecystectomy: A Prospective Randomized Controlled Study
Brief Title: Effects of Intraoperative Warming Methods on Hematologic Inflammatory Indices in Laparoscopic Cholecystectomy
Acronym: WARM-CHOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erkan Cem ÇELİK, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/657; 2025/2 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Inflammatory Response; Perioperative Hypothermia; Laparoscopic Cholecystectomy; Surgical Stress Response
Keywords: Intraoperative warming; Forced-air warming; Combined warming; Hypothermia prevention; Fluid warming; Hematologic inflammatory indices; Neutrophil-to-lymphocyte ratio (NLR); Platelet-to-lymphocyte ratio (PLR); Systemic immune-inflammation index (SII); Laparoscopic surgery; Cholecystectomy

STUDY DESIGN:
Intervention Model Description: In this prospective, randomized, controlled trial, patients will be equally assigned to four groups:
  Control Group (standard blanket + passive blanket)
  IV Warmer Group (standard care + intravenous fluid warmer)
  External Warmer Group (standard care + external warmer)
  Combined Warmer Group (standard care + intravenous fluid warmer + external warmer)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Other): Patients receive standard intraoperative warming with 38 °C set active warming blanket. Surgical field outside the blanket is covered with passive drapes. No additional warming interventions are applied. (standart care)
  Interventions: Device: Standard Active Warming Blanket
- Intravenous Warmer Group (Active Comparator): All standard procedures performed in the control group are followed. Additionally, all intravenous fluids administered during the operation are warmed to 38°C with a fluid warmer.
  Interventions: Device: Standard Active Warming Blanket; Device: Intravenous Warmer Group
- External Warmer Group (Active Comparator): All standard approaches used in the control group are performed. Additionally, a special drape is placed over the upper extremities and thorax, which is connected to a 3M Bair Hugger 700 Series device and warmed to 38°C.
  Interventions: Device: Standard Active Warming Blanket; Device: External Warmer Group
- Combined Warming Group (Intravenous + External) (Active Comparator): All standard approaches used in the control group are performed. Additionally, intravenous fluids are warmed and an external heating device is applied to the upper extremity/thorax.
  Interventions: Device: Standard Active Warming Blanket; Device: Intravenous Warmer Group; Device: External Warmer Group

INTERVENTIONS:
Device: Standard Active Warming Blanket — An active blanket set at 38°C is used to maintain the patient's body temperature throughout the operation. Body areas outside the surgical field are covered with passive drapes. No supplemental heating is used.
  Other Names: MEDWARM W-300/A 150-MS/A 96116-K4656
Device: Intravenous Warmer Group — All intravenous fluids administered during the operation are administered via a fluid warming device at 38°C. All standard practices continue in the control group.
  Other Names: IV Fluid Warmer; Portable Flotherm QW3 Fluid And Blood Warmer
  Arms: Combined Warming Group (Intravenous + External); Intravenous Warmer Group
Device: External Warmer Group — A special drape is placed over the upper extremities and thorax, and the patient is connected to an external warm air device at 38°C throughout the operation. All standard practices continue in the control group.
  Other Names: External Forced-Air Warming Device; 3M Bair Hugger 700 Series
  Arms: Combined Warming Group (Intravenous + External); External Warmer Group

SUMMARY:
Perioperative hypothermia is a frequent and preventable complication that may cause adverse outcomes such as increased blood loss, impaired coagulation, and delayed recovery. Various active warming techniques are used to maintain normothermia during anesthesia; however, their comparative effects on systemic inflammatory responses remain unclear.

This randomized controlled clinical trial aims to evaluate the effects of different intraoperative warming methods on hematologic inflammatory indices - including neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), and systemic immune-inflammation index (SII) - in patients undergoing elective laparoscopic cholecystectomy under general anesthesia.

A total of eligible adult patients will be randomly assigned into four groups according to the intraoperative warming method applied:

Control Group: No active warming applied.

Forced-Air Warming (FAW) Group: Warming blanket system used throughout surgery.

Fluid Warming (FW) Group: Intravenous fluids warmed to maintain normothermia.

Combined Warming (FAW + FW) Group: Both forced-air and fluid warming applied simultaneously.

Core body temperature and perioperative data will be recorded. Venous blood samples will be obtained preoperatively and 24 hours postoperatively to calculate inflammatory indices.

The primary objective is to determine whether active intraoperative warming techniques modulate postoperative inflammatory markers compared to no warming. Secondary outcomes include intraoperative temperature trends, recovery times, and the incidence of hypothermia-related complications.

The results are expected to identify the most effective warming strategy to minimize inflammation and optimize postoperative recovery in laparoscopic procedures.

DETAILED DESCRIPTION:
Unintended perioperative hypothermia (core temperature <36°C) commonly occurs during laparoscopic surgeries due to anesthesia-induced thermoregulatory impairment, pneumoperitoneum, and cold ambient conditions. Even mild decreases in body temperature can impair coagulation, delay drug metabolism, and alter immune function. Maintaining normothermia is therefore critical for improving surgical outcomes.

While both forced-air warming systems and fluid warming devices are routinely used, limited data exist comparing their individual and combined effects on postoperative inflammatory responses. Hematologic inflammatory indices such as NLR, PLR, and SII provide cost-effective and reproducible markers that reflect systemic inflammation and immune balance.

This prospective, randomized, controlled, parallel-group study will be conducted at Atatürk University Faculty of Medicine, Department of Anesthesiology and Reanimation.

Eligible participants are adult patients (aged 18-65 years, ASA I-II) scheduled for elective laparoscopic cholecystectomy under general anesthesia. Patients with infection, chronic inflammatory disease, hematologic disorder, or those converted to open surgery will be excluded.

Participants will be randomly assigned to one of four groups:

Group C (Control): No active warming; standard passive insulation only.

Group FAW (Forced-Air Warming): Forced-air warming blanket applied from induction until the end of surgery.

Group FW (Fluid Warming): Intravenous fluids administered through a warming device.

Group CF (Combined Warming): Both forced-air warming and fluid warming used together.

Standardized anesthesia induction and maintenance protocols will be followed for all patients. Core temperature will be continuously monitored via nasopharyngeal probe. Temperature, hemodynamic parameters, and perioperative variables will be recorded at fixed intervals.

Blood samples will be obtained at two time points - preoperatively and at 24 hours postoperatively - for complete blood count analysis. The inflammatory indices (NLR, PLR, SII) will be calculated and compared among groups.

Primary Outcome:

Postoperative change in hematologic inflammatory indices [(neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), and systemic immune-inflammation index (SII)].

Secondary Outcomes:

Intraoperative temperature maintenance, recovery characteristics, and hypothermia-related adverse events.

Statistical analyses will be performed using SPSS. Continuous variables will be expressed as mean ± SD or median (IQR) and analyzed using ANOVA or Kruskal-Wallis test, as appropriate. Categorical data will be compared using Chi-square or Fisher's exact test. A p-value <0.05 will be considered statistically significant.

This study seeks to clarify whether intraoperative thermal management strategies influence the systemic inflammatory response, potentially guiding clinicians toward the most effective warming method to enhance recovery and minimize postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic cholecystectomy.
* ASA (American Society of Anesthesiologists) physical status I-III.
* Age between 18 and 65 years.
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* ASA IV-V patients.
* Emergency surgery requirement.
* Preoperative fever (>38.0 °C) or hypothermia (<36.0 °C).
* Operation duration <60 minutes or >180 minutes.
* Endocrine/metabolic disorders affecting body temperature (e.g., moderate-severe thyroid dysfunction, pheochromocytoma, severe dysautonomia, malnutrition).
* Active infection/sepsis or systemic infection within past 2 weeks.
* Chronic immunosuppressive therapy (e.g., ≥10 mg/day prednisolone equivalent ≥2 weeks or biological agents in the past month).
* Hematologic disorders (e.g., leukemia, aplastic anemia, myeloproliferative disorders) or abnormal blood counts (platelet <100 ×10⁹/L, leukocyte <3 ×10⁹/L).
* Active malignancy or ongoing chemotherapy/radiotherapy in last 3 months.
* Severe organ failure (Child-Pugh C liver, eGFR <30 mL/min/1.73 m² or dialysis, NYHA III-IV heart failure, GOLD III-IV COPD).
* Coagulopathy or uncontrolled antithrombotic therapy.
* Pregnancy or lactation.
* Conversion from laparoscopic to open surgery.
* Non-adherence to assigned warming protocol.
* Inability to place esophageal temperature probe or unreliable temperature monitoring.
* Intraoperative hemodynamic instability requiring prolonged vasopressor support or blood transfusion.
* Missing or incomplete preoperative or postoperative CBC preventing calculation of inflammatory indices.
* Withdrawal of consent or loss to follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative Core Body Temperature | Intraoperative, measured continuously and recorded at the end of surgery (1 time point)
  Core body temperature will be continuously monitored via esophageal probe throughout laparoscopic cholecystectomy. The primary outcome is the mean core temperature at the end of surgery, comparing the four intraoperative warming strategies (Control, IV warming, External warming, Combined IV + External warming).

SECONDARY OUTCOMES:
Systemic Immune-Inflammation Index (SII) | Preoperative baseline, postoperative 1 hour, and postoperative 24 hours
  SII will be calculated using neutrophil, lymphocyte, and platelet counts from complete blood counts to assess systemic inflammatory response.
Neutrophil-to-Lymphocyte Ratio (NLR) | Preoperative baseline, postoperative 1 hour, and postoperative 24 hours
  NLR will be calculated from complete blood counts to evaluate the balance between acute inflammation and immune function.
Platelet-to-Lymphocyte Ratio (PLR) | Preoperative baseline, postoperative 1 hour, and postoperative 24 hours
  PLR will be calculated from platelet and lymphocyte counts to assess postoperative inflammatory and thrombotic response.
Lymphocyte-to-Monocyte Ratio (LMR) | Preoperative baseline, postoperative 1 hour, and postoperative 24 hours
  LMR will be calculated from lymphocyte and monocyte counts to evaluate immune regulation and inflammatory balance after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Erkan Cem Çelik, doctor, Principal Investigator — Ataturk University Department of Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data (demographics, perioperative temperature, hematologic inflammatory indices) will be made available upon reasonable request to qualified researchers after publication of the primary study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data and supporting documents will be available starting 6 months after publication of the primary study results, for a period of 5 years.
Access Criteria: Qualified researchers affiliated with recognized academic or clinical institutions may request access to the de-identified dataset and supporting documents via email to the corresponding author. Requests will be reviewed for scientific validity and compliance with ethical standards, and data will be shared under a data use agreement.

REFERENCES:
- [Result] Wang J, Bi Y, Ma J, He Y, Liu B. Association of Preoperative Neutrophil-to-Lymphocyte Ratio with Postoperative Acute Kidney Injury and Mortality Following Major Noncardiac Surgeries. World J Surg. 2023 Apr;47(4):948-961. doi: 10.1007/s00268-022-06878-2. Epub 2023 Jan 21. PMID 36681771
- [Result] Jiao Y, Zhang X, Liu M, Sun Y, Ma Z, Gu X, Gu W, Zhu W. Systemic immune-inflammation index within the first postoperative hour as a predictor of severe postoperative complications in upper abdominal surgery: a retrospective single-center study. BMC Gastroenterol. 2022 Aug 27;22(1):403. doi: 10.1186/s12876-022-02482-9. PMID 36030214
- [Result] Gao Y, Guo W, Cai S, Zhang F, Shao F, Zhang G, Liu T, Tan F, Li N, Xue Q, Gao S, He J. Systemic immune-inflammation index (SII) is useful to predict survival outcomes in patients with surgically resected esophageal squamous cell carcinoma. J Cancer. 2019 Jun 2;10(14):3188-3196. doi: 10.7150/jca.30281. eCollection 2019. PMID 31289589
- [Result] Xu H, Wang Z, Guan X, Lu Y, Malone DC, Salmon JW, Ma A, Tang W. Safety of intraoperative hypothermia for patients: meta-analyses of randomized controlled trials and observational studies. BMC Anesthesiol. 2020 Aug 15;20(1):202. doi: 10.1186/s12871-020-01065-z. PMID 32799802
- [Result] Zheng W, Huang B, Bao L, Wang J, Jin J. Comparing warming strategies to reduce hypothermia and shivering in elderly abdominal or pelvic surgery patients: a network meta-analysis. Sci Rep. 2025 Jul 1;15(1):22356. doi: 10.1038/s41598-025-04644-7. PMID 40595941
- [Result] Ji N, Wang J, Li X, Shang Y. Strategies for perioperative hypothermia management: advances in warming techniques and clinical implications: a narrative review. BMC Surg. 2024 Dec 30;24(1):425. doi: 10.1186/s12893-024-02729-0. PMID 39736577
- [Result] McSwain J. Perioperative hypothermia: Causes, consequences and treatment. World Journal of Anesthesiology. 11/27 2015;4:58. doi:10.5313/wja.v4.i3.58
- [Result] Rauch S, Miller C, Brauer A, Wallner B, Bock M, Paal P. Perioperative Hypothermia-A Narrative Review. Int J Environ Res Public Health. 2021 Aug 19;18(16):8749. doi: 10.3390/ijerph18168749. PMID 34444504
- [Result] Reynolds L, Beckmann J, Kurz A. Perioperative complications of hypothermia. Best Pract Res Clin Anaesthesiol. 2008 Dec;22(4):645-57. doi: 10.1016/j.bpa.2008.07.005. PMID 19137808
- [Result] Ruetzler K, Kurz A. Consequences of perioperative hypothermia. Handb Clin Neurol. 2018;157:687-697. doi: 10.1016/B978-0-444-64074-1.00041-0. PMID 30459033